CLINICAL TRIAL: NCT05672914
Title: Intervening to Promote Tobacco Cessation Following Psychiatric Hospitalization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Ascension Seton Shoal Creek (Unknown); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Richard A. Brown, Research Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002552; RP220203 (Other Grant/Funding Number: Cancer Prevention & Research Institute of Texas)
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet-based Sustained Care (Experimental): Intervention to support sustained smoking cessation.
  Interventions: Behavioral: Tablet-based sustained care
- Usual Care (No Intervention): Standard hospital care: : A brief (5-10 min.) tobacco education session from a hospital nurse, along with educational materials about quitting and a quitline brochure.

INTERVENTIONS:
Behavioral: Tablet-based sustained care — A tablet-based motivational-interviewing intervention, tailored specifically to smokers with psychiatric disorders, to motivate the use of evidence-based tobacco treatment and cessation in cigarette smokers upon discharge from an inpatient psychiatric hospitalization. In addition, participants will receive standard hospital tobacco care (see Usual Care Arm).
  Arms: Tablet-based Sustained Care

SUMMARY:
Cigarette smoking is the leading cause of death and disability in the United States. People with psychiatric disorders consume almost half (44.3%) of all cigarettes smoked in the U.S. and have life spans more than 20 years shorter than the general population. Effective quit smoking treatments for people with psychiatric disorders are sorely needed.

When patients are hospitalized for a psychiatric disorder, they are not allowed to smoke. This enforced period of no smoking creates what professionals call "a teachable moment". It provides an excellent opportunity to discuss the prospect of staying quit once the individual leaves the hospital.

In ongoing research, the investigators have developed and tested a Sustained Care quit smoking intervention for smokers engaged in a psychiatric hospitalization. The intervention includes: 1) a professionally-led, motivational counseling session to encourage quitting smoking and increase awareness about available quit smoking resources, 2) a referral to the Texas Tobacco Quitline for phone-based, quit smoking counseling, and 3) an offer of 8 weeks of nicotine patches after leaving the hospital. Findings from a recently completed clinical trial provide strong support for this Sustained Care intervention.

Aims in the current project are to develop and test a tablet computer-based, motivational counseling intervention that does not require a trained professional counselor. The goal is to conduct a clinical trial to demonstrate the effectiveness of this tablet-based, Sustained Care intervention for smokers engaged in psychiatric hospitalization. As before, the same quit smoking resources (Quitline and nicotine patches) will be provided upon hospital discharge. If successful, next steps will involve plans to implement this quit smoking intervention in psychiatric hospitals throughout Texas, in order to reduce the burden caused by tobacco-related cancers among the citizens of Texas.

DETAILED DESCRIPTION:
Cigarette smoking is the leading cause of death in the U.S., resulting in over 480,000 deaths annually. Individuals with any mental illness constitute 18.9% of the U.S. adult population and are estimated to consume almost half (44.3%) of all cigarettes smoked in the U.S. Indeed, individuals with psychiatric disorders smoke cigarettes at disproportionately higher rates and bear an especially large proportion of the tobacco morbidity and mortality burden, with life spans more than 20 years shorter than the general population. People with mental disorders are at significantly elevated risk of malignancies of the brain and central nervous system and respiratory system, including cancers of the lung and bronchus, likely due to cigarette smoking. Yet smokers in inpatient psychiatric settings are rarely encouraged to quit smoking or provided referrals for cessation treatment on discharge, despite growing evidence that smoking cessation may improve psychiatric symptoms long-term and that many smokers with psychiatric disorders want to quit smoking.

Given the disproportionately high rates of smoking and related cancer morbidity and mortality among those with psychiatric disorders, the integration of effective smoking cessation interventions into psychiatric treatment settings is a public health priority. As no tobacco use is allowed on psychiatric hospital units and smoking patterns are disrupted, the inpatient setting in particular offers an ideal opportunity to initiate smoking cessation by capitalizing on abstinence already achieved during hospitalization. This clinical trial attempts to capitalize upon this largely underutilized "teachable moment" by framing a cessation effort as a continuation of what has already begun, i.e., continued movement toward total abstinence.

It was demonstrated, in a randomized controlled trial (RCT) of 342 adult smokers receiving inpatient psychiatric care, that an in-person, motivational interviewing (MI)-based, Sustained Care (SusC) intervention (including tobacco quitline referral and nicotine patches) vs. Usual Care (UC) resulted in significantly increased smoking cessation treatment utilization and significantly higher rates of confirmed smoking abstinence at 6-months post-hospital discharge. While successful in increasing treatment utilization and confirmed abstinence rates after discharge, this in-person, 40-minute MI intervention would be challenging to implement broadly in psychiatric hospitals across the State of Texas. Inexpensive and readily disseminable options are needed.

The investigators plan to accomplish the objectives of this application by pursuing the following three specific aims. First, to develop a tablet-based (iPad) intervention (named "Tablet-delivered Sustained Care Smoking Cessation Intervention or "T-SusC") intended to motivate the use of evidence-based tobacco treatment and cessation in cigarette smokers upon discharge from an inpatient psychiatric hospitalization. Second, to conduct a Phase III efficacy trial, comparing the effects of T-SusC to Usual Care (UC). We hypothesize that: 2a) T-SusC (vs. UC) will result in higher rates of confirmed 7-day point prevalence abstinence at 1-, 3- and 6-months post-hospital discharge, and 2b) T-SusC (vs. UC) will result in higher rates of utilization of tobacco quitline counseling and smoking cessation medication. Third, to examine potential mechanisms underlying intervention effects. We hypothesize that: 3a) pre-post intervention increases in concerns about smoking and motivation to quit smoking, decreases in concerns about quitting smoking exacerbating psychiatric symptoms and greater satisfaction with intervention content will mediate efficacy and 2b) utilization rates of tobacco quitline engagement and cessation medication use will mediate efficacy. Finally, the effect of T-SusC (vs. UC) on psychiatric symptoms over the course of the 6-month follow-up period will be examined.

The rationale for the proposed research is demonstrated by findings from the prior RCT, showing that many smokers in psychiatric treatment are interested in quitting smoking, and armed with the knowledge that quitting smoking does not jeopardize psychiatric treatment and may improve psychiatric symptoms in the long run, can be motivated to engage in smoking cessation counseling and medication use with good success. This project is expected to result in the development of a brief, cost-effective tablet-based (iPad) MI intervention that will produce increased rates of smoking cessation and increased utilization of tobacco quitline and cessation medication following psychiatric inpatient treatment. These results are expected to have an important positive impact that will move the field closer to the long-term goal of dissemination and integration of the T-SusC into inpatient psychiatric treatment programs throughout Texas, to motivate tobacco cessation in psychiatric patients who smoke.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients above the age of 18 capable of providing informed consent
* Current smoker (at least 5 cigarettes/day when not hospitalized)
* Willing and able to provide informed consent, attend all study visits, and comply with the protocol

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score < 24
* Current diagnosis of dementia or other cognitive impairment that would limit study participation
* Inability to provide consent for study participation due to his/her inability to demonstrate an understanding of study procedures
* Current diagnosis of a (non-nicotine) substance use disorder requiring detoxification
* No access to or inability to communicate by phone, or no stable mailing address
* Planned discharge to institutional care (e.g., nursing home, long-term rehabilitation, jail, etc.)
* Medical contraindication to nicotine patch use
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | 1, 3, and 6 months after hospital discharge
  Binomial outcome of continued smoking abstinence vs. relapse modeled over time and controlling for gender and magnitude of initial nicotine dependence

SECONDARY OUTCOMES:
Number of quit attempts | First month following hospital discharge
  Count of attempts to quit smoking

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brown, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- Ascension Shoal Creek, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No